CLINICAL TRIAL: NCT00915967
Title: Pilot Project: Prevention of Neurosurgical Wound Infections
Brief Title: Prevention of Neurosurgical Wound Infections
Acronym: POWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kim J. Burchiel, Kim J. Burchiel, MD / John Raaf Professor and Chairman, Department of Neurological Surgery, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_5170
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-01

CONDITIONS: Surgical Wound Infections
Keywords: Infection; Vancomycin; Neurosurgery; Stimulator; Pump; Deep Brain Stimulation; Intrathecal Pump
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — Vancomycin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin (Experimental): Subjects in the experimental group will receive Vancomycin injected directly into the wound pocket.
  Interventions: Drug: Vancomycin
- Saline (Placebo Comparator): Subjects in the saline group will receive a Saline injection directly into the wound pocket.
  Interventions: Drug: Placebo (Saline Solution)

INTERVENTIONS:
Drug: Vancomycin — Subjects randomized to the vancomycin group will receive an injection (up to 10 mL) of 5 mg/mL vancomycin administered directly into the wound with a blunt needle following watertight fascial closure.
  Arms: Vancomycin
Drug: Placebo (Saline Solution) — Subjects randomized to the saline group will receive an injection (up to 10 mL) of saline solution directly into the wound following watertight fascial closure.
  Arms: Saline

SUMMARY:
The goal of this study is to determine whether injecting the antibiotic vancomycin directly into surgical wounds can decrease the rate of infection following implantation of neurosurgical devices.

ELIGIBILITY:
Inclusion Criteria:

* deep brain stimulators (DBS)
* spinal cord stimulators (SCS)
* motor cortex stimulators (MCS)
* vagus nerve stimulators (VNS)
* peripheral nerve stimulators (PNS)

Exclusion Criteria:

* allergies to vancomycin
* immunocompromise or taking immunosuppressant drugs
* currently taking aminoglycoside antibiotics, such as amikacin, gentamicin, neomycin, streptomycin or tobramycin
* diagnosed renal failure
* currently undergoing chemotherapy
* pregnancy
* non-english speakers
* unable to return for follow-up, or unable to be contacted by telephone

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-05-13 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim J Burchiel, MD, Principal Investigator — Department of Neurological Surgery, Oregon Health & Science University; Valerie C Anderson, PhD, MCR, Principal Investigator — Department of Neurological Surgery, Oregon Health & Science University; Stephen T Magill, PhD, Principal Investigator — School of Medicine, Oregon Health & Science University
Locations (1):
- University Hospital, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Miller JP, Acar F, Burchiel KJ. Significant reduction in stereotactic and functional neurosurgical hardware infection after local neomycin/polymyxin application. J Neurosurg. 2009 Feb;110(2):247-50. doi: 10.3171/2008.6.17605. PMID 19263587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 214 subjects signed consent. 198 subjects were enrolled.
Period: Overall Study
Arm/Group | Vancomycin | Saline
Started | 98 | 100
Completed | 97 | 98
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | Saline | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Least Squares Mean (Inter-Quartile Range); unit: Years] | 63 [55 to 71] | 64 [54 to 74] | 63.5 [54 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 58 | 63 | 121
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 98 | 100 | 198

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infection That Requires Removal of the Neurosurgical Device
Description: The primary outcome was infection that required removal of the implanted device within 6 months of surgery. At our institution all patients with evidence of hardware infection have the entire stimulation/pump system removed. Subjects were either seen in clinic or reached by telephone more than 6 months after surgery and assessed for whether they had had infection requiring hardware removal or any superficial infection requiring additional post-operative antibiotics.
Time Frame: Six months post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Saline
Number analyzed (Participants) | 98 | 100
Participants | 97 | 98

ADVERSE EVENTS:
Time Frame: 6 months
Description: The study aimed to determine whether retrospectively observed decrease in infection rate could be attributed to the addition of local antibiotics A prospective, randomized, double-blind, placebo-controlled pilot study comparing standard antibiotic prophylaxis with addition of local intrawound injection of vancomycin or placebo, was designed.
  Study Procedures were standard of care, risk was minimal
Arm/Group | Vancomycin | Saline
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/100
Other Adverse Events (participants affected / at risk) | 2/98 | 5/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin (N=98) | Saline (N=100)
Infection (Surgical and medical procedures) | 2 (2) | 5 (5) — Wound Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No